CLINICAL TRIAL: NCT04658628
Title: Brain Imaging Biomarkers for Response to Spinal Cord Stimulation in Patients With Chronic Low Back Pain
Status: Recruiting | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Evangelia C. Tsolaki, MSc, PhD, Principal Investigator, University of California, Los Angeles
Other Study IDs: IRB#20-001870
Record Dates: First submitted 2020-11-24; First posted 2020-12-08 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Chronic Low-back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
In this protocol, "Brain imaging biomarkers for response to Spinal Cord Stimulation in patients with chronic low back pain," the investigators plan to perform brain mapping studies in 42 patients who are undergoing spinal cord stimulation (SCS) for chronic low back pain (CLBP) as part of the participants normal clinical care during a 2-year period. This imagining study is completed for research purposes. There is no standard of care imaging for the participants. This study requires two visits in total. During the baseline visit, participants will undergo imaging acquisition protocol and corresponding assessments. Participants will have another follow-up visit (potentially remotely) for final assessments two weeks after the SCS treatment. The objective of the study is to investigate potential imaging biomarkers that can predict response to the SCS treatment. Specifically, the investigators hypothesize that the connectivity of a certain region of the brain (specifically the subgenual cingulate) prior to SCS may serve as a possible pre-operative imaging-based biomarker on response to SCS. The findings of the study may further enhance investigators understanding of the connectivity between brain areas that are critical to the therapeutic response to SCS in CLBP patients and that can be used as a putative biomarker to select patients who may respond to SCS.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 21 years of age at time of consent
* Subject has been recommended to undergo an SCS trial for chronic back with or without leg pain by their pain management physician
* Chronic low back pain as defined by persistent low back pain despite prior treatments that continues for 12 weeks or longer
* Subject signs a valid, Institutional Review Board (IRB)-approved informed consent form (ICF) provided

Exclusion Criteria:

* Subject is a woman who is not using adequate contraception, is pregnant or breastfeeding or intends to become pregnant during the course of the study
* Subject has previously undergone a spinal cord stimulation trial or is already implanted with an active implantable device(s) to treat their pain (Implantable Pulse Generators (IPGs), implantable drug pump, etc.) or pacemaker or implantable cardiac defibrillator
* Subject is currently abusing alcohol or illicit drugs
* Contraindications to MRIs or the need for recurrent body MRIs
* Presence of cardiac pacemakers/defibrillators, implanted medication pumps, intra-cardiac lines, any intracranial implants (e.g., aneurysm clip, shunt, cochlear implant, electrodes) or other implanted stimulators

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults recommended to undergo an SCS trial for chronic back with or without leg pain by their pain management physician
Sampling Method: Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2021-01-22 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Change in VAS | Baseline and 2 weeks
  The visual analog scale for pain is a continuous horizontal scale of length 100mm with the extremes of pain expressed on either end (left = no pain, right = worst pain).
Change in HAMD-17 | Baseline and 2 weeks
  The HAMD-17 is a 17-item scale that evaluates depressed mood, vegetative and cognitive symptoms of depression, and comorbid anxiety symptoms. The HAMD-17 was one of the first rating scales developed to quantify the severity of depressive symptomatology. First introduced by Max Hamilton in 1960, it has since become the most widely used and accepted outcome measure for evaluating depression severity. It provides ratings on current Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) symptoms of depression, with the exception of hypersomnia, increased appetite, and concentration/indecision. The HAMD-17 was designed to be administered by a trained clinician using a semi-structured clinical interview. The 17-items are rated on either a 5-point (0-4) or a 3-point (0-2) scale.
Change in MPQ | Baseline and 2 weeks
  The Short-Form McGill Pain Questionnaire (SF-MPQ) is used for the measurement of pain. The measure is calculated by summing the point values for responses to 15 questions. Questions 1-11 deal with the sensory dimension of pain (i.e., the quality of the pain). Questions 12-15 deal with the affective dimension of pain (i.e., how the pain affects you). Subscores for the sensory and affective dimensions are calculated, in addition to a total McGill Pain Score. Higher scores generally correspond to an worsened subjective experience of pain.
Change in PASS | Baseline and 2 weeks
  The PASS--20 measures fear and anxiety responses specific to pain. It includes four subscales that reflect aspects of avoidance behavior, cognitive anxiety, fear, and physiological anxiety. All items are rated on a scale from 0 (never) to 5 (always).

CONTACTS AND LOCATIONS:
Locations (1):
- University of California Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No